CLINICAL TRIAL: NCT04432831
Title: A Multicenter, Open-Label Extension Study to Evaluate the Long-Term Safety and Tolerability of Faricimab in Patients With Diabetic Macular Edema
Brief Title: A Study to Evaluate the Long-Term Safety and Tolerability of Faricimab in Participants With Diabetic Macular Edema
Acronym: Rhone-X
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR41987; 2020-000402-29 (EudraCT Number)
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Masking Description: The first 16 weeks of this study will be a masked period (to transition from the multi-arm parent studies) during which participants may receive either faricimab or sham injection. Participants and physicians will be masked only to the faricimab treatment interval. After the Week 16 treatment procedure, this study will follow an open-label design. The BCVA examiner will remain masked for the duration of this long-term extension study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Faricimab PTI (Experimental)
  Interventions: Drug: Faricimab; Other: Sham Procedure

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered by intravitreal (IVT) injection into the study eye according to the personalized treatment interval (PTI) dosing regimen.
  Other Names: RO6867461; RG7716
Other: Sham Procedure — The sham is a procedure that mimics an IVT injection and involves the blunt end of an empty syringe (without a needle) being pressed against the anesthetized eye. The sham procedure will be administered to participants as appropriate during the first 16 weeks of this study in order to maintain the masking of the initial faricimab PTI.

SUMMARY:
This is a multicenter long-term extension study designed to evaluate the long-term safety and tolerability of faricimab administered by intravitreal (IVT) injection at a personalized treatment interval (PTI) to participants who enrolled in and completed one of the two Phase III studies, GR40349 (NCT03622580) or GR40398 (NCT03622593), also referred to as the parent studies.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in and completion of Study GR40349 (NCT03622580) or GR40398 (NCT03622593), without study or study drug discontinuation
* Ability to comply with the study protocol, in the investigator's judgment
* For women of childbearing potential: agreement to remain abstinent or use acceptable contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 3 months after the final dose of study treatment

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within 3 months after the final intravitreal injection of faricimab
* Presence of other ocular diseases that give reasonable suspicion of a disease or condition that contraindicates the use of faricimab, that might affect interpretation of the results of the study or that renders the patient at high risk for treatment complications
* Presence of other diseases, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of faricimab and that might affect interpretation of the results of the study or that renders the patient at high risk of treatment complications
* History of a severe allergic reaction or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of the faricimab injections, study treatment procedure, dilating drops, or any of the anesthetic and antimicrobial preparations used by a patient during the study
* Requirement for continuous use of any medications or treatments indicated as prohibited therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1479 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (320):
- United States (119):
  - Barnet Dulaney Perkins Eye Center, Mesa, Arizona
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - California Retina Consultants., Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Retinal Diagnostic Center, Campbell, California
  - The Retina Partners, Encino, California
  - Eye Medical Center, Fresno, California
  - Retina Consultants of Orange County, Fullerton, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - East Bay Retina Consultants, Oakland, California
  - Southern CA Desert Retina Cons, Palm Desert, California
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retina Consultants, San Diego, Poway, California
  - Retina Consultants of Southern California, Redlands, California
  - Retinal Consultants Med Group, Sacramento, California
  - West Coast Retina Medical Group, San Francisco, California
  - Orange County Retina Med Group, Santa Ana, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants - Santa Maria, Santa Maria, California
  - Bay Area Retina Associates, Walnut Creek, California
  - University of Colorado; dept of ophthalmology, Aurora, Colorado
  - Retina Consultants of Southern, Colorado Springs, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Rand Eye, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Care Specialists, Palm Beach Gardens, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Fort Lauderdale Eye Institute, Plantation, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Assoc, Tallahassee, Florida
  - Retina Associates of Florida, LLC, Tampa, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Prairie Eye & LASIK Center / Prairie Retina Center, Springfield, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Retina Associates, Lenexa, Kansas
  - Vitreo-Retinal Consultants, Wichita, Kansas
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Med; Wilmer Eye Inst, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina PC, Hagerstown, Maryland
  - Retina Specialists, Towson, Maryland
  - Tufts Medical Center; Ophthalmology, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Beetham Eye Institute, Joslin Diabetes Center, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Associated Retinal Consultants, Grand Rapids, Michigan
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Assoc Retinal Consultants PC, Royal Oak, Michigan
  - Associated Retinal Consultants, P.C., Traverse City, Michigan
  - VitreoRetinal Surgery, PLLC.; DBA Retina Consultants of Minnesota, Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - NJRetina, Edison, New Jersey
  - Retinal & Ophthalmic Cons PC, Northfield, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Capital Region Retina, Albany, New York
  - Long Is. Vitreoretinal Consult, Great Neck, New York
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - Retina Vit Surgeons/Central NY, Liverpool, New York
  - New York University, New York, New York
  - Ophthalmic Cons of Long Island, Oceanside, New York
  - Retina Associates of Western New York, Rochester, New York
  - Island Retina, Shirley, New York
  - The Retina Consultants, Slingerlands, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Char Eye Ear &Throat Assoc, Charlotte, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - Wake Forest Baptist Health Eye Centre, Winston-Salem, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - Cleveland Clinic Foundation; Cole Eye Institute, Cleveland, Ohio
  - The Ohio State University Havener Eye Institute, Columbus, Ohio
  - Midwest Retina, Dublin, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Retina Northwest, Portland, Oregon
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Mid-Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Consultants Of Carolina, Greenville, South Carolina
  - Charleston Neuroscience Inst, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina & Vitreous of Texas, Bellaire, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Texas Retina Associates, Dallas, Texas
  - Valley Retina Institute P.A., Harlingen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Eye Care Assoc of East Texas, Tyler, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Associates of Utah, PLLC, Salt Lake City, Utah
  - University of Utah; Division of Gastroenterology/Hepatology, Salt Lake City, Utah
  - Uni of Vermont Medical Center;, Burlington, Vermont
  - Univ of Virginia Ophthalmology, Charlottesville, Virginia
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Kapoor Institute, Norfolk, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - West Virginia University Eye Institute, Morgantown, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Argentina (6):
  - Fundacion Zambrano, CABA
  - Oftalmos, Capital Federal
  - Oftar, Mendoza
  - Centro Oftalmólogos Especialistas, Rosario
  - Grupo Laser Vision, Rosario
  - Organizacion Medica de Investigacion, San Nicolás
- Australia (7):
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Sydney Retina Clinic and Day Surgery, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Austria (4):
  - LKH-Univ.Klinikum Graz; Universitäts-Augenklinik, Graz
  - Kepler Universitätskliniken GmbH - Med Campus III; Abt. für Augenheilkunde, Linz
  - Medizinische Universität Wien; Universitätsklinik für Augenheilkunde und Optometrie, Vienna
  - Hanusch Krankenhaus; Abteilung für Augenkrankheiten mit Augen-Tagesklinik, Vienna
- Brazil (9):
  - Hospital de Olhos de Aparecida - HOA, Aparecida de Goiânia, Goiás
  - Centro Brasileiro de Cirurgia, Goiânia, Goiás
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Botelho Hospital da Visao, Blumenau, Santa Catarina
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP*X; Oftalmologia, São Paulo, São Paulo
  - CEMAPE - Centro Médico, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
  - Hosp de Olhos de Sorocaba, Sorocaba, São Paulo
- Bulgaria (4):
  - Medical Center for Eye Health ? Focus Ltd, Sofia
  - Pentagram Eye Hospital (Medical Center "Pentagram"), Sofia
  - Spec. Ophth. Hospital for Active Treatment- Academic Pashev, Sofia
  - Specialized Hospital for Active Treatment of Eye Diseases Zora, Sofia
- Canada (7):
  - Calgary Retina Consultants, Calgary, Alberta
  - QEII - HSC Department of Ophthalmology, Halifax, Nova Scotia
  - Ivey Eye Institute, London, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - St. Michael's Hospital; Department of Ophthalmology, Toronto, Ontario
  - University Health Network Toronto Western Hospital, Toronto, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
- Czechia (5):
  - FN Hradec Králové, Ocní klinika; Ophthalmology clinic, Hradec Králové
  - Faculty Hospital Ostrava; Ophthalmology clinic, Ostrava
  - Faculty Hospital Kralovske Vinohrady; Ophthalmology clinic, Prague
  - AXON Clinical, Prague
  - Nemocnice Sokolov, Sokolov
- Denmark (2):
  - Aalborg Universitetshospital; Øjenafdelingen, Aalborg
  - Sjællands Universitetshospital, Roskilde; Øjenafdelingen, Roskilde
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux Hopital Pellegrin, Bordeaux
  - Chi De Creteil; Ophtalmologie, Créteil
  - Pole Vision Val d'Ouest; Ophtalmologie, Écully
  - CHU Nantes - Hôtel Dieu; Ophthalmology, Nantes
  - Hopital Lariboisiere; Ophtalmologie, Paris
  - Centres Ophtalmologique St Exupéry; Ophtalmologie, Saint-Cyr-sur-Loire
- Germany (10):
  - Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Augenheilkunde, Dresden
  - Universitätsklinikum Freiburg, Klinik für Augenheilkunde, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Klinik für Augenheilkunde, Hanover
  - Universitätsklinikum des Saarlandes; Klinik für Augenheilkunde, Homburg/Saar
  - Universitätsklinikum Magdeburg A.ö.R., Universitätsaugenklinik, Magdeburg
  - LMU Klinikum der Universität, Augenklinik, München
  - Klinikum rechts der Isar der TU München; Augenklinik, München
  - Augenabteilung am St. Franziskus-Hospital, Münster
  - Universitätsklinikum Münster; Augenheilkunde, Münster
  - Universitätsklinikum Würzburg, Augenklinik und Poliklinik, Würzburg
- Hong Kong (2):
  - Queen Mary Hospital; Department of Ophthalmology, Hong Kong
  - Hong Kong Eye Hospital; CUHK Eye Centre, Mong Kok
- Hungary (10):
  - Eszak-Pesti Centrumkorhaz - Honvedkorhaz; Szemeszet, Budapest
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Baleseti Kozpont, Szemeszet KR, Budapest
  - Semmelweis Egyetem Szemészeti Vizsgálóhely, Budapest
  - Bajcsy-Zsilinszky Hospital, Budapest
  - Budapest Retina Associates Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont; Szemeszeti Klinika, Debrecen
  - Ganglion Medial Center, Pécs
  - Szegedi Tudományegyetem ÁOK; Department of Ophtalmology, Szeged
  - Markusovszky Egyetemi Oktatokorhaz ; SZEMESZET; Intezeti Gyogyszertar, Szombathely
  - Zala Megyei Kórház; SZEMESZET, Zalaegerszeg
- Israel (5):
  - Rambam Medical Center; Opthalmology, Haifa
  - Hadassah MC; Ophtalmology, Jerusalem
  - Rabin MC; Ophtalmology, Petah Tikva
  - Kaplan Medical Center; Ophtalmology, Rehovot
  - Tel Aviv Sourasky MC; Ophtalmology, Tel Aviv
- Italy (8):
  - Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia-Presidio Ospedaliero Britannico, Rome, Lazio
  - UNIVERSITA' DEGLI STUDI DI GENOVA - Di.N.O.G.;CLINICA OCULISTICA, Genoa, Liguria
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico-Clinica Regina Elena;U.O.C Oculistica, Milan, Lombardy
  - Irccs Ospedale San Raffaele;U.O. Oculistica, Milan, Lombardy
  - Azienda Ospedaliero-Universitaria Careggi; S.O.D. Oculistica, Florence, Tuscany
  - Nuovo Ospedale S. Chiara - A.O.U.P Presidio Ospedaliero di Cisanello; U.O. Oculistica Universitaria, Pisa, Tuscany
  - Azienda Ospedaliera di Perugia Ospedale S. Maria Della Misericordia; Clinica Oculistica, Perugia, Umbria
  - Ospedale Classificato Equiparato Sacro Cuore ? Don Calabria; Presso Ufficio Cassa, Negrar - Verona, Veneto
- Japan (23):
  - Sugita Eye Hospital, Aichi
  - Nagoya University Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Aichi Medical University Hospital, Aichi
  - Toho University Sakura Medical Center, Chiba
  - Hayashi Eye Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Asahikawa Medical University Hospital, Hokkaido
  - Hyogo Prefectural Amagasaki General Medical Center (Hyogo AGMC), Hyōgo
  - Kozawa eye hospital and diabetes center, Ibaraki
  - Ideta Eye Hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - Mie University Hospital, Mie
  - University of Miyazaki Hospital, Miyazaki
  - Nara Medical University Hospital, Nara
  - Kitano Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - National Defense Medical College Hospital, Saitama
  - Shiga University Of Medical Science Hospital, Shiga
  - Tokyo Women's Medical University, Tokyo
  - Kyorin University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
- Mexico (4):
  - Centro Oftalmológico Mira, S.C, Del. Cuauhtemoc, Mexico CITY (federal District)
  - Macula Retina Consultores, México, Mexico CITY (federal District)
  - Hospital de la Ceguera APEC, México, Mexico CITY (federal District)
  - Instituto de la retina del Bajio, Querétaro City, Querétaro
- Peru (3):
  - Mácula D&T, Lima
  - TG Laser Oftalmica, Lima
  - Oftalmolaser, Lima
- Poland (16):
  - Szpital sw. Lukasza, Bielsko-Biala
  - Specjalistyczny Osrodek Okulistyczny Oculomedica, Bydgoszcz
  - OFTALMIKA Sp. z o.o, Bydgoszcz
  - Szpital Specjalistyczny nr 1; Oddzial Okulistyki, Bytom
  - Dobry Wzrok Sp Z O O, Gdansk
  - Optimum Profesorskie Centrum Okulistyki, Gdansk
  - Poradnia Okulistyczna i Salon Optyczny w Gliwicach- PRYZMAT, Gliwice
  - Gabinet Okulistyczny Prof Edward Wylegala, Katowice
  - Centrum Medyczne UNO-MED, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie Oddzia? Kliniczny Okulistyki i Onkologii Okulistycznej, Krakow
  - Optomed Sp. z o.o., Rybnik
  - Osrodek Chirurgii Oka prof. Zagorskiego Rzeszow, Rzeszów
  - Kliniczny Szpital Wojewodzki nr 1 im. F. Chopina; Klinika Okulistyki, Rzeszów
  - Caminomed, Tarnowskie Góry
  - Centrum Zdrowia MDM, Warsaw
  - SPEKTRUM Osrodek Okulistyki Klinicznej, Wroclaw
- Portugal (4):
  - Hospital de Braga; Servico de Oftalmologia, Braga
  - AIBILI - Association for Innovation and Biomedical Research on Light, Coimbra
  - Espaco Medico Coimbra, Coimbra
  - Hospital de Santa Maria; Servico de Oftalmologia, Lisbon
- Russia (7):
  - Clinic Optimed, Ufa, Bashkortostan Republic
  - Intersec Research and Technology Complex ?Eye Microsurgery? n.a. S.N. Fyodorov; Cheboksary Branch, Cheboksary, Mariy-El Republic
  - FSBI ?Scientific Research Institute of Eye Diseases? of Russian Academy of medical Sciences, Moscow, Moscow Oblast
  - Medical Military Academy n.a S.M.Kirov, Saint Petersburg, Sankt-Peterburg
  - Clinics of Eye Diseases, LLC, Kazan', Tatarstan Republic
  - ?Intersec. Research and Technology Complex ?Eye Microsurgery? n a Fyodorov Irkutsk branch, Irkutsk
  - ?Intersec Research and Technology Complex Eye Microsurgery n a Fyodorov Novosibirsk Branch, Novosibirsk
- Singapore (3):
  - National University Hospital; Ophthalmology Department, Singapore
  - Singapore Eye Research Institute, Singapore
  - Tan Tock Seng Hospital; Ophthalmology Department, Singapore
- Slovakia (3):
  - Nemocnica s poliklinikou Trebišov, a.s., Trebišov
  - Fakultna nemocnica Trencin Ocna klinika, Trenčín
  - Fakultna nemocnica s poliklinikou Zilina; Ocne oddelenie, Žilina
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (18):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Instituto Oftalmologico Gomez Ulla; Servicio de Oftalmologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario de Gran Canaria; Servicio de oftalmologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Clinica Universitaria de Navarra; Servicio de Oftalmologia, Pamplona, Navarre
  - Complejo Hospitalario de Navarra; Servicio de oftalmologia, Pamplona, Navarre
  - Instituto Oftalmologico Fernandez Vega; Servicio de oftalmologia, Oviedo, Principality of Asturias
  - Oftalvist Valencia, Burjassot, Valencia
  - Complejo Hospitalario Universitario Albacete; Servicio de oftalmologia, Albacete
  - VISSUM Instituto Oftalmológico de Alicante, Alicante
  - Centro de Oftalmologia Barraquer; Servicio Oftalmologia, Barcelona
  - Hospital dos de maig; servicio de oftalmologia, Barcelona
  - Hospital Clinic de Barcelona; Consultas Externas Oftalmologia, Barcelona
  - Hospital de Santa Creu I Sant Pau; Servicio de Oftalmologia, Barcelona
  - Clinica Baviera; Servicio Oftalmologia, Madrid
  - Fisabio-Ofalmologia Medica; Servicio de Oftalmología, Valencia
  - Hospital Universitario Rio Hortega; Servicio de Oftalmologia, Valladolid
- Vista Klinik Ophthalmologische Klinik, Binningen, Switzerland
- Taiwan (3):
  - Taipei Veterans General Hospital; Ophthalmology, Taipei
  - Chang Gung Medical Foundation - Linkou; Ophthalmology, Taoyuan District
  - National Taiwan University Hospital; Ophthalmology, Zhongzheng Dist.
- Thailand (3):
  - King Chulalongkorn Memorial Hospital; Ophthalmology Department, Bangkok
  - Rajavithi Hospital; Ophthalmology Department, Bangkok
  - Maharaj Nakorn ChiangMai Hospital; Ophthalmology Department, Chiang Mai
- Turkey (Türkiye) (7):
  - Hacettepe University Medical Faculty; Department of Ophthalmology, Ankara
  - Ankara University Medical Faculty; Department of Ophthalmology, Ankara
  - Ankara Baskent University Medical Faculty; Department of Ophthalmology, Ankara
  - Beyoglu Goz Training and Research Hospital; Department Of Ophthalmology, Istanbul
  - Ege University Medical Faculty; Department of Ophthalmology, Izmir
  - Kocaeli Üniversitesi T?p Fakültesi; Department of Ophthalmology, Kocaeli
  - Selcuk University Faculty of Medicine; Department Of Ophthalmology, Konya
- United Kingdom (16):
  - Hillingdon Hospital, Uxbridge, Middx
  - James Paget University Hospitals NHS Foundation Trust, Great Yarmouth, Norfolk
  - Belfast Health and Social Care Trust, ROYAL VICTORIA HOSPITAL, Belfast
  - Bradford Royal Infirmary, Bradford
  - East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Frimley Park Hospital, Frimley
  - Gloucestershire Hospitals NHS Foundation Trust, Gloucester
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital; St Paul's Clinical Eye Research Centre, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Royal Free Hospital, London
  - Kings College Hospital, London
  - Manchester Royal Eye Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University Hospital Southampton NHS Foundation Trust; Southampton Eye Unit, Southampton
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Result] Sheth VS, Schlottmann P, Lai TYY, Abreu F, Chang A, Eter N, Gibson K, Hu AY, Korobelnik JF, Kotak A, Kotecha A, O'Leary OE, Pearce I, Sim DA, Sun JK, Tang Y, Khanani AM. Four-Year Outcomes of Faricimab in Diabetic Macular Edema: Results From the RHONE-X Extension Trial. Ophthalmology. 2026 Jan 12:S0161-6420(26)00004-7. doi: 10.1016/j.ophtha.2026.01.001. Online ahead of print. PMID 41534798

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1479 patients were enrolled, but 5 participants in total were excluded from the analysis populations because of Good Clinical Practice (GCP) non-compliance at a single site.
Groups:
- Faricimab PTI (Prior Faricimab Q8W): This analysis group includes participants who were previously randomized to Arm A (faricimab 6 mg Q8W) in one of the parent studies, GR40349 (NCT03622580) and GR40398 (NCT03622593), and then enrolled in this extension study to receive faricimab 6 mg by IVT injection according to the personalized treatment interval (PTI) dosing regimen.
- Faricimab PTI (Prior Faricimab PTI): This analysis group includes participants who were previously randomized to Arm B (faricimab 6 mg PTI) in one of the parent studies, GR40349 (NCT03622580) and GR40398 (NCT03622593), and then enrolled in this extension study to receive faricimab 6 mg by IVT injection according to the personalized treatment interval (PTI) dosing regimen.
- Faricimab PTI (Prior Aflibercept Q8W): This analysis group includes participants who were previously randomized to Arm C (aflibercept 2 mg Q8W) in one of the parent studies, GR40349 (NCT03622580) and GR40398 (NCT03622593), and then enrolled in this extension study to receive faricimab 6 mg by IVT injection according to the personalized treatment interval (PTI) dosing regimen.
Period: Overall Study
Arm/Group | Faricimab PTI (Prior Faricimab Q8W) | Faricimab PTI (Prior Faricimab PTI) | Faricimab PTI (Prior Aflibercept Q8W)
Started | 493 | 506 | 475
Received at Least One Dose of Study Drug (Safety-Evaluable Population) | 491 | 500 | 473
Completed | 405 | 407 | 392
Not Completed | 88 | 99 | 83
Not completed — Withdrawal by Subject | 24 | 28 | 21
Not completed — Death | 23 | 23 | 17
Not completed — Lost to Follow-up | 15 | 15 | 12
Not completed — Final End of Study Visit Not Completed | 10 | 11 | 7
Not completed — Reason Not Specified | 7 | 11 | 9
Not completed — Adverse Event | 7 | 7 | 7
Not completed — Physician Decision | 1 | 3 | 6
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: A total of 1479 patients consented to enroll in RHONE-X once they completed the parent studies. However, the baseline analysis population includes a total of 1474 participants because 5 participants were excluded from all analyses as an outcome of the GCP non-compliance identified at one of the clinical trial sites.
Groups:
- Total: Total of all reporting groups
Arm/Group | Faricimab PTI (Prior Faricimab Q8W) | Faricimab PTI (Prior Faricimab PTI) | Faricimab PTI (Prior Aflibercept Q8W) | Total
Number analyzed (Participants) | 493 | 506 | 475 | 1474
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (9.9) | 64.0 (9.8) | 63.5 (9.4) | 63.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 184 | 205 | 580
  Male | 302 | 322 | 270 | 894
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 87 | 79 | 234
  Not Hispanic or Latino | 415 | 408 | 386 | 1209
  Unknown or Not Reported | 10 | 11 | 10 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 4 | 13
  Asian | 54 | 52 | 45 | 151
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Black or African American | 27 | 32 | 25 | 84
  White | 392 | 406 | 389 | 1187
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 13 | 12 | 11 | 36

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular Adverse Events in the Study Eye, With Severity Determined According to Adverse Event Severity Grading Scale
Description: This is an analysis of participants with at least one ocular adverse event (AE) that occurred in the study eye. Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of the seriousness, severity (e.g., mild, moderate, or severe intensity), and causality for each AE. AEs of special interest (AESI) included the following: Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, are associated with severe intraocular inflammation (IOI), or require surgical or medical intervention to prevent permanent loss of sight; suspected transmission of an infectious agent by the study drug; and, cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From the day of the first dose of faricimab until the end of the study (up to 108 weeks)
Population: The Safety-Evaluable Population included all participants who enrolled in this long-term extension (LTE) study and received at least one dose of faricimab in the study eye during the LTE. A total of 10 participants who were enrolled in the study but did not receive treatment with faricimab were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Faricimab PTI (Prior Faricimab Q8W) | Faricimab PTI (Prior Faricimab PTI) | Faricimab PTI (Prior Aflibercept Q8W)
Number analyzed (Participants) | 491 | 500 | 473
Participants
  Any Adverse Event (AE), Any Severity | 219 | 188 | 197
  AE by Severity: Mild | 119 | 109 | 109
  AE by Severity: Moderate | 74 | 66 | 74
  AE by Severity: Severe | 20 | 10 | 12
  AE by Severity: Missing | 6 | 3 | 2
  Serious Adverse Event (SAE) | 31 | 15 | 26
  AE Leading to Withdrawal from Study Treatment | 3 | 0 | 6
  Treatment-related AE | 10 | 10 | 11
  Treatment-related SAE | 0 | 1 | 1
  Any AE of Special Interest (AESI) | 30 | 14 | 24
  AESI: Drop in Visual Acuity Score ≥30 Letters | 23 | 10 | 20
  AESI: Associated with Severe IOI | 1 | 1 | 1
  AESI: Intervention Required to Prevent Permanent Vision Loss | 6 | 3 | 3
  AESI: Suspected Transmission of Infectious Agent by Study Drug | 0 | 0 | 0

2. Primary Outcome: Incidence of Ocular Adverse Events in the Fellow Eye
Description: This is an analysis of participants with at least one ocular adverse event (AE) that occurred in the fellow eye (i.e., non-study eye). Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of the seriousness, severity, and causality for each AE. AEs of special interest (AESI) included the following: Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, are associated with severe intraocular inflammation (IOI), or require surgical or medical intervention to prevent permanent loss of sight; suspected transmission of an infectious agent by the study drug; and, cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From the day of the first dose of faricimab until the end of the study (up to 108 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Faricimab PTI (Prior Faricimab Q8W) | Faricimab PTI (Prior Faricimab PTI) | Faricimab PTI (Prior Aflibercept Q8W)
Number analyzed (Participants) | 491 | 500 | 473
Participants
  Any Adverse Event (AE) | 186 | 185 | 179
  Serious Adverse Event (SAE) | 16 | 17 | 15
  Any AE of Special Interest (AESI) | 13 | 16 | 14
  AESI: Drop in Visual Acuity Score ≥30 Letters | 6 | 9 | 10
  AESI: Associated with Severe IOI | 0 | 1 | 1
  AESI: Intervention Required to Prevent Permanent Vision Loss | 7 | 6 | 4
  AESI: Suspected Transmission of Infectious Agent by Study Drug | 0 | 0 | 0

3. Primary Outcome: Incidence and Severity of Non-Ocular Adverse Events, With Severity Determined According to Adverse Event Severity Grading Scale
Description: This is an analysis of participants with at least one non-ocular (systemic) adverse event (AE). Investigators sought information on AEs at each contact with the participants. All AEs were recorded and the investigator made an assessment of the seriousness, severity (e.g., mild, moderate, or severe intensity), and causality for each AE. AEs of special interest (AESI) included the following: Sight-threatening AEs that cause a drop in visual acuity (VA) score ≥30 letters lasting more than 1 hour, are associated with severe intraocular inflammation (IOI), or require surgical or medical intervention to prevent permanent loss of sight; suspected transmission of an infectious agent by the study drug; and, cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law.
Time Frame: From the day of the first dose of faricimab until the end of the study (up to 108 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Faricimab PTI (Prior Faricimab Q8W) | Faricimab PTI (Prior Faricimab PTI) | Faricimab PTI (Prior Aflibercept Q8W)
Number analyzed (Participants) | 491 | 500 | 473
Participants
  Any Adverse Event (AE), Any Severity | 317 | 295 | 297
  AE by Severity: Mild | 91 | 94 | 97
  AE by Severity: Moderate | 124 | 124 | 115
  AE by Severity: Severe | 102 | 77 | 85
  Serious Adverse Event (SAE) | 122 | 100 | 112
  AE Leading to Withdrawal from Study Treatment | 2 | 7 | 4
  Any AE of Special Interest (AESI) | 0 | 0 | 1
  AESI: Drop in Visual Acuity Score ≥30 Letters | 0 | 0 | 1
  AESI: Elevated ALT or AST with Either Elevated Bilirubin or Clinical Jaundice | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the day of the first dose of faricimab until the end of the study (up to 108 weeks)
Description: For All-Cause Mortality: all participants enrolled in the study. For AEs: the Safety-Evaluable Population included all participant who enrolled and received at least one dose of faricimab during the study. For ocular AEs, the number of participants and events reported per term are specified to have occurred in the study eye or the fellow eye.
Arm/Group | Faricimab PTI (Prior Faricimab Q8W) | Faricimab PTI (Prior Faricimab PTI) | Faricimab PTI (Prior Aflibercept Q8W)
All-Cause Mortality (participants affected / at risk) | 23/493 | 23/506 | 17/475
Serious Adverse Events (participants affected / at risk) | 158/491 | 124/500 | 134/473
Other Adverse Events (participants affected / at risk) | 233/491 | 213/500 | 219/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faricimab PTI (Prior Faricimab Q8W) (N=491) | Faricimab PTI (Prior Faricimab PTI) (N=500) | Faricimab PTI (Prior Aflibercept Q8W) (N=473)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 3 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 4 (4) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 4 (6)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Cardiac discomfort (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (4) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (9) | 3 (4) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 6 (6) | 5 (5) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 9 (9) | 3 (3) | 8 (8)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — SAEs occurred in the fellow eye
Cataract (Eye disorders) | 11 (11) | 8 (8) | 15 (15) — SAEs occurred in the study eye
Cataract cortical (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — SAEs occurred in the fellow eye
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — SAEs occurred in the study eye
Diabetic retinal oedema (Eye disorders) | 7 (8) | 0 (0) | 2 (2) — SAEs occurred in the study eye
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — SAEs occurred in the study eye
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — SAEs occurred in the study eye
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — SAEs occurred in the study eye
Iridocele (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — SAEs occurred in the study eye
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — SAEs occurred in the study eye
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — SAEs occurred in the fellow eye
Posterior capsule opacification (Eye disorders) | 2 (2) | 0 (0) | 0 (0) — SAEs occurred in the study eye
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1) | 2 (2) — SAEs occurred in the study eye
Retinal detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0) — SAEs occurred in the study eye
Retinal neovascularisation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — SAEs occurred in the fellow eye
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — SAEs occurred in the study eye
Retinal vein occlusion (Eye disorders) | 2 (2) | 1 (1) | 0 (0) — SAEs occurred in the study eye
Rhegmatogenous retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — SAEs occurred in the study eye
Tractional retinal detachment (Eye disorders) | 2 (2) | 0 (0) | 0 (0) — SAEs occurred in the fellow eye
Uveitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) — SAEs occurred in the study eye
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 2 (2) — SAEs occurred in the study eye
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral mucosal hypertrophy (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Death (General disorders) | 3 (3) | 5 (5) | 2 (2)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0)
Organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 2 (2)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 10 (10) | 9 (9) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 2 (2) | 3 (3)
Cellulitis (Infections and infestations) | 3 (3) | 4 (4) | 6 (6)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Diabetic gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) — SAEs occurred in the study eye
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 2 (2) | 3 (4)
Gastroenteritis norovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infected skin ulcer (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 7 (7) | 0 (0) | 2 (3)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 7 (7) | 4 (4) | 0 (0)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 8 (9) | 3 (4)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 2 (2) | 4 (4)
Septic endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Systemic bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cataract traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — SAEs occurred the study eye
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — SAEs occurred in the fellow eye
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — SAEs occurred the study eye
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ocular procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — SAEs occurred in the fellow eye
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural constipation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — SAEs occurred in the fellow eye
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ammonia increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glycosylated haemoglobin abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) — SAEs occurred in the fellow eye
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Precancerous cells present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 3 (3) | 10 (10)
Encephalomalacia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — SAEs occurred in the fellow eye
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1)
Vertebral artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (9) | 5 (5) | 5 (7)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (2)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1) | 0 (0)
Renal haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Orchitis noninfective (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cellulite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 3 (3)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (2) | 3 (3) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 6 (6) | 0 (0) — SAEs occurred in the fellow eye
Diabetic retinal oedema (Eye disorders) | 1 (1) | 1 (1) | 2 (2) — SAEs occurred in the fellow eye
Diabetic retinopathy (Eye disorders) | 2 (2) | 3 (3) | 2 (2) — SAEs occurred in the fellow eye
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 2 (2) — SAEs occurred in the fellow eye
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — SAEs occurred in the fellow eye
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — SAEs occurred in the fellow eye
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — SAEs occurred in the fellow eye
Vitreous haemorrhage (Eye disorders) | 4 (4) | 3 (3) | 6 (6) — SAEs occurred in the fellow eye
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) — SAEs occurred in the fellow eye
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faricimab PTI (Prior Faricimab Q8W) (N=491) | Faricimab PTI (Prior Faricimab PTI) (N=500) | Faricimab PTI (Prior Aflibercept Q8W) (N=473)
Cataract (Eye disorders) | 65 (65) | 60 (60) | 63 (63) — AEs occurred in the study eye
Diabetic retinal oedema (Eye disorders) | 22 (22) | 27 (31) | 24 (27) — AEs occurred in the fellow eye
Posterior capsule opacification (Eye disorders) | 16 (17) | 17 (17) | 14 (14) — AEs occurred in the study eye
COVID-19 (Infections and infestations) | 63 (70) | 49 (50) | 46 (49)
Conjunctival haemorrhage (Eye disorders) | 16 (17) | 9 (9) | 5 (5) — AEs occurred in the study eye
Diabetic retinopathy (Eye disorders) | 17 (17) | 8 (8) | 12 (12) — AEs occurred in the fellow eye
Vitreous detachment (Eye disorders) | 16 (16) | 12 (12) | 6 (6) — AEs occurred in the study eye
Vitreous floaters (Eye disorders) | 16 (18) | 7 (7) | 8 (8) — AEs occurred in the study eye
Nasopharyngitis (Infections and infestations) | 18 (21) | 12 (12) | 23 (27)
Urinary tract infection (Infections and infestations) | 16 (19) | 15 (17) | 16 (18)
Intraocular pressure increased (Investigations) | 16 (20) | 12 (15) | 12 (13) — AEs occurred in the study eye
Hypertension (Vascular disorders) | 18 (18) | 20 (20) | 23 (24)
Cataract (Eye disorders) | 56 (56) | 41 (41) | 51 (52) — AEs occurred in the fellow eye
Posterior capsule opacification (Eye disorders) | 13 (14) | 20 (20) | 13 (13) — AEs occurred in the fellow eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT04432831/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT04432831/SAP_001.pdf